CLINICAL TRIAL: NCT01310205
Title: An Extension of Study SCI-SCV-HCV-P2-001: Long-Term FU in Subj Who Opt for Retreatment With Pegylated Interferon and Ribavirin After Completing Treatment in a Phase 2 Study and Have Relapsed After at Least 44 Weeks Tx With Peg-IFN and RBV.
Brief Title: Extension Study SCI-SCV-HCV-P2-001: Long-Term FU in Subj Who Opt for Retreatment With Peg-INF and RBV After Completing Treatment in HCV
Status: Completed | Type: Observational
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SCI-SCV-HCV-P2-001-Extension
Record Dates: First submitted 2011-03-04; First posted 2011-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Genotype 1; relapsers; non cirrhotic; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — golotimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatitis C treatment: This is an extension of ongoing study SCI-SCV-HCV-P2-001. Subjects will be invited to participate in this extension study if they complete treatment in study SCI-SCV-HCV-P2-001 and are eligible for retreatment with peg-IFN and RBV
  Interventions: Drug: SCV-07
- non cirrhotic subjects: This is an extension of ongoing study SCI-SCV-HCV-P2-001. Subjects will be invited to participate in this extension study if they complete treatment in study SCI-SCV-HCV-P2-001 and are eligible for retreatment with peg-IFN and RBV
  Interventions: Drug: SCV-07

INTERVENTIONS:
Drug: SCV-07 — This is an extension of ongoing study SCI-SCV-HCV-P2-001. Subjects will be invited to participate in this extension study if they complete treatment in study SCI-SCV-HCV-P2-001 and are eligible for retreatment with peg-IFN and RBV

SUMMARY:
This is an extension of ongoing study SCI-SCV-HCV-P2-001 in which subjects will be invited to participate in this extension study if they complete treatment in study SCI-SCV-HCV-P2-001 and are eligible for retreatment with peg-IFN and RBV.

DETAILED DESCRIPTION:
In this extension study, subjects will be asked to give permission to share their HCV RNA viral load test results, obtained from local laboratories, at the different time points and will also be asked to give permission to share their SOC dosing information (peg-IFN and RBV). As no SCV-07 treatment, procedures, or assessments will be required during this extension study, no related safety information will be collected.

The study will last up to 72 weeks after subjects complete treatment on study SCI-SCV-HCV-P2-001 and begin retreatment with peg-IFN and RBV.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who satisfy all of the following criteria may be enrolled into the study:

Subjects must be able to understand and sign an ICF approved by the investigator's institutional review board (IRB) for this study; must have completed treatment on study SCI-SCV-HCV-P2-001; and must, in the judgment of the investigators, be able to benefit from retreatment per current SOC (peg-IFN and RBV).

Exclusion Criteria:

* Subjects who satisfy any of the following criteria will not be enrolled into the study:

Subjects who, in the opinion of the investigators, will be unable to tolerate retreatment with peg-IFN and RBV for at least 48 weeks and are at high risk of early treatment discontinuation and plan to participate in another investigational trial prior to providing a final sample for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an extension of ongoing study SCI-SCV-HCV-P2-001. Subjects will be invited to participate in this extension study if they complete treatment in study SCI-SCV-HCV-P2-001 and are eligible for retreatment with peg-IFN and RBV
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Modelska, MD, Study Director — SciClone Pharmaceuticals
Locations (4):
- United States (4):
  - AGMG Clinical Research, Anaheim, California
  - Univ of Louisville Med/Dental Complex, Louisville, Kentucky
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Walter Reed Army Medical Center, Washington, Washington

REFERENCES:
- See also: Sponsor — http://www.sciclone.com